CLINICAL TRIAL: NCT01289938
Title: Pharmacogenetic Factors and Side Effects of Metoclopramide and Diphenhydramine
Acronym: MalD
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: To unsuccessful recruitment of rare UM-genotype. All other planned genotype groups are completed (EM, IM and PM).
Sponsor: Matthias Schwab (Other)
Responsible Party: Sponsor-Investigator, Matthias Schwab, Prof. M.D., University Hospital Tuebingen
Organization: University Hospital Tuebingen (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IKP231; 2008-003778-16 (EudraCT Number)
Record Dates: First submitted 2011-02-02; First posted 2011-02-04 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Drug Metabolism, Poor, CYP2D6-RELATED
Keywords: pharmacokinetic; pharmacogenetic; Metoclopramide; Diphenhydramine; CYP2D6 polymorphisms
MeSH Terms: conditions — Drug Metabolism, Poor, CYP2D6-Related | interventions — Diphenhydramine; Metoclopramide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metoclopramide (Active Comparator): Metoclopramide treatment
  Interventions: Drug: Metoclopramide
- Diphenhydramine (Active Comparator): Diphenhydramine treatment
  Interventions: Drug: Diphenhydramine

INTERVENTIONS:
Drug: Diphenhydramine — Diphenhydramine 50 mg oral once
  Other Names: DPH
  Arms: Diphenhydramine
Drug: Metoclopramide — 10 mg i.v. metoclopramide once
  Other Names: MCP
  Arms: Metoclopramide

SUMMARY:
Pharmacokinetic of Metoclopramide (MCP) in correlation to polymorphisms of CYP2D6 and Dopamine-D2-Receptor. Pharmacokinetic of Diphenhydramine (DPH) in correlation to polymorphisms of CYP2D6

ELIGIBILITY:
Inclusion Criteria:

* BMI 20 - 27kg/m2
* Caucasians
* Healthy volunteers

Exclusion Criteria:

* Pregnancy/lactation period
* Drug allergy
* Acute and chronic diseases
* Taking medication
* Abuse of drugs, alcohol etc.
* Smoker

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2009-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Area under curve of metoclopramide (MCP) | 0,5, 1, 1,5, 2, 3, 4, 6, 8, 12, 24, 34, 48, 72 hours
  Pharmacokinetic of MCP at following time points:
  0,5, 1, 1,5, 2, 3, 4, 6, 8, 12, 24, 34, 48, 72 hours after drug application
Area under curve of diphenhydramine(DPH) | 0,5, 1, 1,5, 2, 3, 4, 6, 8, 12, 24, 34, 48, 72 hours
  Pharmacokinetics of DPH at following time points:
  0,5, 1, 1,5, 2, 3, 4, 6, 8, 12, 24, 34, 48, 72 hours after drug application

SECONDARY OUTCOMES:
Cmax of metoclopramide | 0,5, 1, 1,5, 2, 3, 4, 6, 8, 12, 24, 34, 48, 72 hours
  Cmax of metoclopramide at following time points:
  0,5, 1, 1,5, 2, 3, 4, 6, 8, 12, 24, 34, 48, 72 hours after drug application
Tmax of metoclopramide | 0,5, 1, 1,5, 2, 3, 4, 6, 8, 12, 24, 34, 48, 72 hours
  Tmax of metoclopramide at following time points:
  0,5, 1, 1,5, 2, 3, 4, 6, 8, 12, 24, 34, 48, 72 hours after drug application
Cmax of diphenhydramine | 0,5, 1, 1,5, 2, 3, 4, 6, 8, 12, 24, 34, 48, 72 hours
  Cmax of diphenhydramine at the following time points:
  0,5, 1, 1,5, 2, 3, 4, 6, 8, 12, 24, 34, 48, 72 hours after drug application
Tmax of diphenhydramine | 0,5, 1, 1,5, 2, 3, 4, 6, 8, 12, 24, 34, 48, 72 hours
  Tmax of diphenhydramine at the following time points:
  0,5, 1, 1,5, 2, 3, 4, 6, 8, 12, 24, 34, 48, 72 hours after drug application

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Schwab, MD, Principal Investigator — UKT
Locations (1):
- Abteilung Klinische Pharmakologie, UKT Tübingen, Tübingen, Baden-Wurttemberg, Germany

REFERENCES:
- [Background] Kirchheiner J, Seeringer A. Clinical implications of pharmacogenetics of cytochrome P450 drug metabolizing enzymes. Biochim Biophys Acta. 2007 Mar;1770(3):489-94. doi: 10.1016/j.bbagen.2006.09.019. Epub 2006 Oct 4. PMID 17113714
- [Background] Schroth W, Antoniadou L, Fritz P, Schwab M, Muerdter T, Zanger UM, Simon W, Eichelbaum M, Brauch H. Breast cancer treatment outcome with adjuvant tamoxifen relative to patient CYP2D6 and CYP2C19 genotypes. J Clin Oncol. 2007 Nov 20;25(33):5187-93. doi: 10.1200/JCO.2007.12.2705. PMID 18024866